CLINICAL TRIAL: NCT00238940
Title: A One-year, Randomized, Open Label, Parallel Group Study to Investigate the Safety and the Effect of Enteric-coated Mycophenolate Sodium (EC-MPS) in Combination With Either Full Dose or Reduced Dose Cyclosporine Microemulsion in de Novo Kidney Transplant Recipients
Brief Title: Extension Study of Enteric-coated Mycophenolate Sodium in Combination With Full Dose or Reduced Dose Cyclosporine Microemulsion in Patients With de Novo Kidney Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405DE01E1
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
This extension study is considered to allow patients being treated with EC-MPS to collect further information on the long-term safety of this drug.

ELIGIBILITY:
Inclusion/ Exclusion criteria

- All patients who completed study CERL080A2405-DE01 and who are willing to continue treatment with EC-MPS.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Efficacy based on level of serum creatinine and calculated creatinine clearance 6 months post transplantation.

SECONDARY OUTCOMES:
Efficacy based on the level of serum creatinine and calculated creatinine clearance 12 months post transplantation.
Safety and tolerability of enteric-coated mycophenolate sodium at 6 and 12 months post transplantation
Pharmacokinetics enteric coated mycophenolate sodium in a randomized subgroup
Efficacy based on the incidence of biopsy-proven acute rejection, graft loss or death 6 and 12 months post transplantation.
Efficacy based on the incidence of biopsy-proven acute rejection at 6 and 12 months post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis